CLINICAL TRIAL: NCT03359343
Title: Computer-aided Classification of Colorectal Polyp by Using Linked Colour Imaging
Brief Title: Computer-assisted Diagnosis System Based on Linked Colour Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 307-LCI-CAD
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Polyp; Linked Color Imaging; Computer-aided Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- experts: In this group, two experts distinguish a set of polyps on LCI images as adenoma or non-adenoma.
- non-experts: In this group, two non-experts distinguish the set of polyps(the same to experts group) on LCI images as adenoma or non-adenoma.
- Computer-aided diagnosis system: In this group, a newly developed computer-aided diagnosis system will be used to distinguish a set of polyps as adenoma or non-adenoma.

SUMMARY:
Linked color imaging (LCI)，a new endoscopy modality, creates clear and bright images by using short wavelength narrow band laser light. LCI can make red area appear redder and white areas appear whiter. Thus, it may be possible to distinguish adenoma and non-adenoma polyps based on color evaluation of LCI images. This study aimed to assess the correlation between histology results and LCI images. Moreover, the investigators conducted a pilot study to explore the clinical potential of LCI to distinguish adenoma and non-adenoma polyps and the accuracy of an automatic computer-aided diagnosis system using LCI imagine to predict histology polyps when compared to human experts physicians.

DETAILED DESCRIPTION:
This study consists of a retrospective analysis and a pilot study. In the retrospective study, the investigators tried to find out an correlation between LCI images and histology results for polyp lesions. And a computer-aided analysis of the images was conducted to demonstrate the correlation objectively. Thereafter,a pilot study was performed to explore whether the previous correlation could be easily learned to distinguish adenoma and non-adenoma polyps by comparing the results of experts diagnosis of LCI image and non-experts. Also, in the pilot study, the investigators assessed the accuracy of an automate histology diagnosis method for polyp LCI images using the computer-aided system when compared to human experts physicians. Throughout the entire research, histology results are regarded as gold standard.

ELIGIBILITY:
Inclusion Criteria:

- at least one polyp found during colonoscopy examination.

Exclusion Criteria:

- poor quality of bowel preparation which impedes histology evaluation; previous resection of colon; inflammatory bowel disease; familiar adenomatous polyposis; Peutz-Jeghers syndrome or other polyposis syndrome.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients undergoing colonoscopy
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
LCI accuracy | June 1, 2018
  the accuracy between a novel developed computer-aided diagnosis system and human experts physicians o distinguish adenoma polyps and non-adenoma polyps based on LCI image.

SECONDARY OUTCOMES:
the short learning curve | June 1, 2018
  the accuracy between experts and non-experts to distinguish adenoma polyps and non-adenoma polyps based on LCI image was compared to explore whether LCI method is of an shorter learning curve.
the correlation | June 1, 2018
  the correlation between LCI image and histology results were retrospectively explored

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, Study Director — Department of gastroenterology, Affiliated Hospital to Academy of Military Medical Sciences.
Locations (2):
- China (2):
  - Affiliated Hospital to Academy of Military Medical Sciences, Beijing, Beijing Municipality
  - Department of Gastroenterology, Affilited Hospital to Academy of Military Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fukuda H, Miura Y, Hayashi Y, Takezawa T, Ino Y, Okada M, Osawa H, Lefor AK, Yamamoto H. Linked color imaging technology facilitates early detection of flat gastric cancers. Clin J Gastroenterol. 2015 Dec;8(6):385-9. doi: 10.1007/s12328-015-0612-9. Epub 2015 Nov 11. PMID 26560036
- [Background] Sun X, Dong T, Bi Y, Min M, Shen W, Xu Y, Liu Y. Linked color imaging application for improving the endoscopic diagnosis accuracy: a pilot study. Sci Rep. 2016 Sep 19;6:33473. doi: 10.1038/srep33473. PMID 27641243
- [Background] Dohi O, Yagi N, Onozawa Y, Kimura-Tsuchiya R, Majima A, Kitaichi T, Horii Y, Suzuki K, Tomie A, Okayama T, Yoshida N, Kamada K, Katada K, Uchiyama K, Ishikawa T, Takagi T, Handa O, Konishi H, Naito Y, Itoh Y. Linked color imaging improves endoscopic diagnosis of active Helicobacter pylori infection. Endosc Int Open. 2016 Jul;4(7):E800-5. doi: 10.1055/s-0042-109049. PMID 27556101